CLINICAL TRIAL: NCT00541567
Title: A Placebo-Controlled, Randomized, Double-Blind, Parallel Arm, Multicenter, Dose-Ranging Phase IIb Trial to Assess Glycemic and Weight Loss Efficacy and Safety of BMS-646256 in Overweight and Obese Patients With Type 2 Diabetes Inadequately Controlled by Diet and Exercise Only or With Metformin or Sulfonylurea Monotherapy
Brief Title: BMS-646256 in Obese and Overweight Type 2 Diabetics
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Veronika von Hahn, Solvay Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S319.2.002; EudraCT No. 2007-005124-32
Record Dates: First submitted 2007-10-09; First posted 2007-10-10 (Estimated); Last update posted 2008-01-09 (Estimated); Status verified 2008-01

CONDITIONS: Obesity and Type 2 Diabetes
Keywords: Wheight management in T2D
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — ibipinabant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Placebo Comparator)
  Interventions: Drug: ibipinabant
- 2 (Experimental)
  Interventions: Drug: ibipinabant
- 3 (Experimental)
  Interventions: Drug: ibipinabant
- 4 (Experimental)
  Interventions: Drug: ibipinabant

INTERVENTIONS:
Drug: ibipinabant — oral, tablet, once daily

SUMMARY:
This is a placebo-controlled, randomized, double-blind, parallel arm, multicenter, dose-ranging phase IIb trial to assess glycemic and weight loss efficacy and safety of BMS-646256 in overweight and obese patients with type 2 diabetes who have been treated with diet and exercise only or with half-maximal or greater metformin (≥1500mg/day) or sulfonylurea monotherapy (stable dose for at least three months), but who remained inadequately controlled (HbA1c >7% and HbA1c<10%).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70 years and BMI ≥27 with type 2 diabetes who have been treated with diet and exercise only or with half maximal or greater metformin or sulfonylurea monotherapy (stable dose for at least three months), but who remained inadequately controlled (HbA1c >7% and HbA1c<10%).

Exclusion Criteria:

* Pregnancy
* Anti-diabetic medications other than baseline metformin or sulfonylurea monotherapy
* History of myocardial infarction in the prior six months/ History of heart failure defined as New York Heart Association Functional Class I, II, III or IV/ History of symptomatic arrhythmia
* Active hepatic disease/ Any documented muscle disease
* History of multiple sclerosis/ Baseline history of tremors, ataxia, anxiety or dizziness
* Seizures within the last year, stroke, and transient ischemic attack/ Known history of schizophrenia, dementia, or bipolar disorder as defined by DSM IV criteria.
* Currently depressed subjects or a CES-D score greater or equal to 16 at the screening visit or at baseline (Day 1)/ History of suicide attempt or ideation
* Previous history of surgical procedures for weight loss (e.g. stomach stapling, bypass)/ Weight loss greater than 5 kg in the prior 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2008-03; Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Absolute change from baseline in body weight (kg) and HbA1c (%) | 26 weeks of double-blind therapy

SECONDARY OUTCOMES:
Waist circumference, fasting glucose and insulin, HOMA analysis, blood lipids (triglycerides, total cholesterol, HDL-C, LDL-C, ApoB) and systolic/ diastolic blood pressure | 52 weeks treatment followed by 20 weeks off-medication period

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals